CLINICAL TRIAL: NCT02830750
Title: A Multi Center Registry of Low- Fluoroscopy Atrial Fibrillation Ablation Using Electroanatomic Mapping Carto
Brief Title: Low Fluoroscopy Afib Ablation Registry
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Beacon Medical Group (Unknown); Brigham and Women's Hospital (Other); Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Responsible Party: Principal Investigator, Gerri O'Riordan, Direcetor of Clinical Resarch. CV Med, Stanford University
Other Study IDs: 35821
Record Dates: First submitted 2016-06-28; First posted 2016-07-13 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Ablation

SUMMARY:
Prospective data collection of patients undergoing Atrial Fibrillation Ablation.

DETAILED DESCRIPTION:
Clinicians who have experience using low dose fluoroscopy including use of Carto Mapping system will consent patients to allow data collection and a 12 month f/up visit to track adverse events. Clinicians will follow a protocol which will be similar to their standard of care for ablations.

ELIGIBILITY:
Inclusion Criteria:

* Patient meets accepted AHA/ACC/HRS guideline indications for catheter ablation of paroxysmal or persistent AF
* First or subsequent ablation procedures may be included
* Age 18-75

Exclusion Criteria:

* Known venous malformations or implanted instrumentation (IVC filter)
* Known PV stenosis
* Unable to provide consent
* H/O mechanical mitral valve replacement (unable to rely on EA mapping only)
* Documented left atrial thrombus
* Prior ASD repair Pregnancy
* NYHA >=3
* EF less than 35%
* CHF within 90 daysRecent MI or coronary revascularization within 90 days
* NOTE: H/O implanted pacemaker or ICD with transvenous leads will NOT be an exclusion criteria, but we will track patients treated with pre-existing transvenous leads with the hypothesis that although fluoroscopy use will be higher in these patients compared to those without leads, but still lower than conventionally treated patients.
* Patients who are undergoing non- standard of care ablations ie, Cyro or FIRM ablations

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have persistant or paroxysmal atrial fibrillation
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2016-04; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Atrial Fibrillation | 12 months
  Determine Atrial Fibrillation burden at 12 month visit by reviewing monitoring systems that capture this data

SECONDARY OUTCOMES:
Fluoroscopic Usage | post operative
  To determine total amount of radiation used at each procedure by estimation of mGy

CONTACTS AND LOCATIONS:
Overall Officials: Chad Brodt, MD PHD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Beacon Medical Group, South Bend, Indiana
  - Brigham's Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No